CLINICAL TRIAL: NCT05001282
Title: Dose Escalation and Expansion Clinical Study to Evaluate the Safety and Efficacy of ELU001 in Subjects Who Have Advanced, Recurrent or Refractory FRα Overexpressing Tumors
Brief Title: A Study to Evaluate ELU001 in Patients With Solid Tumors That Overexpress Folate Receptor Alpha (FRα)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding - no safety issue with Drug; Company Permanently Closed
Sponsor: Elucida Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELU-FRα-1
Record Dates: First submitted 2021-07-14; First posted 2021-08-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma; Endometrial Cancer; Ovary Cancer; Ovary Neoplasm; Ovary Disease; Ovary Metastasis; Ovarian Diseases; Ovarian Cancer Stage; Ovarian Epithelial Cancer; Ovarian Adenocarcinoma; Ovarian Serous Adenocarcinoma; Ovarian Neoplasm Epithelial; Ovarian Cancer Recurrent; Endometrial Diseases; Endometrial Adenocarcinoma; Endometrial Carcinosarcoma; Endometrial Clear Cell Adenocarcinoma; Endometrioid Adenocarcinoma; Endometrial Neoplasms; Endometrial Cancer Recurrent; Endometrioid Tumor; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Folate Receptor Alpha; Carcinomas; Recurrent, Refractory; Folate Receptor alpha moderate expression; Folate Receptor alpha high expression; ELU001; Exatecan; C'Dot; C-Dot; Folic Acid; Payload; Nanoparticle; C'Dot drug conjugate; CDC; Linker; ELU-FRa-1; FOLR1
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Ovarian Diseases; Krukenberg Tumor; Carcinoma, Ovarian Epithelial; Uterine Diseases; Carcinoma, Endometrioid; Fallopian Tube Neoplasms; Carcinoma; Recurrence

STUDY DESIGN:
Intervention Model Description: Dose Escalation Dose Expansion, Simon's 2-stage
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELU001 (Experimental): Dose Escalation: Escalating doses of ELU001 Dose Expansion: Recommended Dose for Expansion (or RP2D)
  Interventions: Drug: ELU001

INTERVENTIONS:
Drug: ELU001 — Folic-acid functionalized C'Dot-Drug-Conjugate (FA-CDC)
  Other Names: FA-CDC

SUMMARY:
This study, ELU- FRα-1, was focused on adult subjects who have advanced, recurrent or refractory folate receptor alpha (FRα) overexpressing tumors considered to be topoisomerase 1 inhibitor-sensitive based on scientific literature, and, in the opinion of the Investigator, have no other meaningful life-prolonging therapy options available.

DETAILED DESCRIPTION:
The study had two parts: Part 1 Dose Escalation Safety Study to identify the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D), and Part 2 Tumor Group Expansion Cohort(s) where specific cancer types will be evaluated for efficacy and safety at the RP2D.

Part 1, subjects with cancer types with a high likelihood of having FRα overexpressing tumors based on historical data, specifically, ovarian, endometrial, colorectal, gastric, gastroesophageal junction, triple negative breast, or non-small cell lung cancers, or cholangiocarcinoma, will be enrolled in a basket clinical study. Retrospective analysis of folate receptor alpha (FRα) expression status will be determined. Part 1 is currently closed for further recruitment.

Part 2 Stage 1 of a Simon's Two-Stage design, tumor group expansion cohorts, each consisting of subjects with cancer types studied as part of the basket in Part 1. Part 2 is closed for recruitment.

ELIGIBILITY:
Key Inclusion Criteria:

Patients must meet the following criteria to enroll in this study:

* Part 1 Documented diagnosis of ovarian cancer, endometrial cancer, colorectal cancer, gastric cancer, gastroesophageal junction cancer, triple negative breast cancer, non-small cell lung cancer, or cholangiocarcinoma
* Part 2 Ovarian Cancer or Endometrial Cancer
* No other meaningful life-prolonging therapy option available
* Must provide archival tumor tissue or a newly obtained tumor biopsy specimen prior to the first dose of ELU001 for folate receptor alpha (FRα) expression analysis. Previous FRα expression test results may be used in certain circumstances
* Adequate organ function
* Measurable disease, or in the absence of measurable disease, non-measurable disease as per Response evaluation criteria in solid tumors (RECIST) v1.1
* Part 1: Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2; Part 2: ECOG performance status of 0 or 1.
* Recovered from previous surgeries
* Agree to highly effective contraception, not to get pregnant, or for men, not father a child during study participation

Key Exclusion Criteria:

Patients who meet any of the following are not eligible to enroll in this study:

* Clinically significant eye disorders
* Taken any treatments that use the protein folate receptor alpha or FRα to work
* Taken any other experimental treatments
* History of significant cardiac issues or other cancers within 3 years.
* Significant anemia, significant neutropenia, or significant thrombocytopenia (e.g., not enough platelets in your blood - platelets held stop bleeding in your body)
* Detectable viral load for HIV (human immunodeficiency virus), hepatitis B or C.
* If you are pregnant.
* Part 1: Cannot have active autoimmune diseases such as rheumatoid arthritis, SLE (systemic lupus erythematosus), ulcerative colitis, Crohn's Disease, MS (multiple sclerosis), ankylosing spondylitis, thyroiditis that require treatments that suppress your immune system.
* Part 1: if your cancer has spread to your brain.
* Part 2: You can have cancer that has spread to your brain but there are exceptions. The cancer in your brain cannot be causing any symptoms, it cannot be larger than 3 cm, there can be no evidence on a scan that shows your brain tissue has shifted from its expected position inside the skull (called "herniation") or be bleeding in the skull or brain itself (called "hemorrhage").

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Part 1 Dose Escalation: The Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of ELU001 for IV infusion in patients with over-expressing Folate Receptor Alpha tumors. | 28 days
  To determine the MTD and/or RP2D of ELU001 in patients with over-expressing Folate Receptor Alpha tumors. When at least 2 out of 6 patients in a given dose-level experience a dose-limiting toxicity (DLT), the dose is considered to have exceeded the MTD. The MTD, therefore, is defined as the previous highest tested dose of ELU001 that did not cause a DLT in the first cycle of treatment. In the event of emerging data during Part 1, the Sponsor may, in consultation with a dose-level safety review group, decide to define a recommended dose for expansion (in for Part 2) (RP2D) instead of the MTD. DLTs are defined as a treatment-emergent adverse event (TEAE) or abnormal laboratory value related to ELU001 treatment that result in a failure to meet the criteria for re-treatment.
Part 2 Dose Expansion: To determine overall response rate (ORR) (complete response [CR] + partial response [PR]) of ELU001 for IV infusion in patients with over-expressing Folate Receptor Alpha tumors, per RECIST v1.1. | First dose of study drug until responses of CR or PR, assessed up to 12 months.
  Percentage of Participants with confirmed objective response as assessed by the investigator and per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 CR is defined as the disappearance of all target or non-target lesions. PR is defined as at least 30 percent (%) decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.

SECONDARY OUTCOMES:
Part 1 Dose Escalation: To determine overall response rate (ORR) (complete response [CR] + partial response [PR]) of ELU001 for IV infusion in patients with over-expressing Folate Receptor Alpha tumors, per RECIST v1.1. | First dose of study drug until responses of CR or PR, assessed up to 12 months.
  Percentage of Participants with confirmed objective response as assessed by the investigator and per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 CR is defined as the disappearance of all target or non-target lesions. PR is defined as at least 30 percent (%) decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.
Part 1 and Part 2: To determine Duration of Response (DOR) of ELU001 for IV infusion in patients with over-expressing Folate Receptor Alpha tumors. | Date of first response (CR or PR) until the date of disease progression or up to 12 months, whichever occurs first.
  Time Measurement: DOR will begin at the date that a response has been identified (stable disease, partial response, or complete response) until the date of progressive disease (PD). PD is defined of at least a 20% increase in the sum of the longest diameters of the target lesions from data of initial response.
Part 1 and Part 2: Number of participants with adverse events as assessed by CTCAE v5.0 Safety Evaluations. | First dose of study drug up to 28 days after the last dose of study drug or up to 12 months, whichever occurs first.
  The number of participants Frequency/severity of abnormalities in vital signs measurements, physical examination findings, changes in clinical laboratory parameters, and incidence of adverse events after taking ELU001.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Mayo Clinic - Phoenix, AZ, Phoenix, Arizona
  - Providence Medical Foundation, Fullerton, California
  - Mayo Clinic - Jacksonville, FL, Jacksonville, Florida
  - D&H Cancer Research Center, Margate, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Mayo Clinic - Rochester, MN, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center - Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - New Experimental Therapeutics of San Antonio (NEXT Oncology), San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No